CLINICAL TRIAL: NCT00468494
Title: Can Blood Glucose Levels During the Perioperative Period Identify a Population at Risk for Hyperglycemia
Brief Title: Can Blood Glucose Levels During the Perioperative Period Identify a Population at Risk for Hyperglycemia?
Status: Completed | Type: Observational
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Other Study IDs: 0120060208
Record Dates: First submitted 2007-04-30; First posted 2007-05-02 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: General Anesthesia; Hyperglycemia
Keywords: non diabetic; catabolic energy state
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Surgery performed during general anesthesia induces a stress effect on the body. Our plan is to identify population at risk of hyperglycemia during perioperative period.

DETAILED DESCRIPTION:
This is a prospective study to define the relationship between time profile of glucose control before, during and after surgery with patient variables, surgical variables and anesthetic variables. Serum glucose levels will be measured preoperatively and then at 30 minute intervals during surgery. Pain score, pain medication and glucose levels will be measured in the post anesthesia recovery room. Subjects will be contacted 2 weeks following the date of surgery to determine the incidence of postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* 18-80 years of age

Exclusion Criteria:

* Known diabetics
* Pregnant patients
* Cardiac surgery patients
* Liver transplant patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: non-diabetic adults undergoing surgery
Sampling Method: Non-Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2006-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
glucose level at specific points | Intraoperatively and in the PACU

SECONDARY OUTCOMES:
pt telephoned to assess for complications | within 2 weeks of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Vasanti Tilak, MD, Principal Investigator — University of Medicine & Dentistry of New Jersey-NJMS
Locations (1):
- University of Medicine & Dentistry of New Jersey, Newark, New Jersey, United States